CLINICAL TRIAL: NCT00962559
Title: Endocrine and Neuropsychological Changes After Aneurismal Subarachnoid Hemorrhage.
Brief Title: Hypopituitarism After Aneurismal Subarachnoid Hemorrhage
Status: Completed | Type: Observational
Sponsor: Universitätsmedizin Mannheim (Other)
Responsible Party: Marcel Seiz, Neurosurgical Department, Universitätsmedizin Mannheim, Theodor-Kutzer-Ufer 1-3, 68167 Mannheim, Germany
Other Study IDs: aSAH and Hypopituitarism 0815
Record Dates: First submitted 2009-08-19; First posted 2009-08-20 (Estimated); Last update posted 2010-02-17 (Estimated); Status verified 2010-02

CONDITIONS: Aneurismal Subarachnoid Hemorrhage; Hypopituitarism; Neuropsychological Deficits
MeSH Terms: conditions — Hypopituitarism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Introduction:

Almost 50% of patients die after aneurismal subarachnoid hemorrhage (aSAH). 30% of the survivors suffer from neurological handicap and need permanent care (Suarez et al.). Even when neurological outcome is good, neuropsychological deficits are frequently observed (Ogden et al., Anderson et al.) The incidence rate of aSAH is almost 8 of 100.000 per year. Due to similar clinical symptoms to patients with hypopituitarism, several studies have analyzed the incidence of hypopituitarism after aSAH. Dysfunction of the anterior pituitary gland was found in up to 47% (Schneider et al.). GH deficiency was demonstrated in almost every fourth patient and an association with poor recovery was postulated. In Germany, the investigators would therefore expect as many as 1200 patients with incident GH deficiency. The KIMS-study is an observational GH-treatment study in adult onset growth hormone deficiency. Within the epidemiological data of KIMS, aSAH is not known as a relevant contributing cause (Brabant et al.). This resembles much of the investigators clinical experience that there is no huge prevalence of hypopituitarism after aSAH.

Objective: Evaluation of the frequency of hypopituitarism and neuropsychological dysfunction of any degree in patients with aSAH in a prospective approach.

Methods:

The investigators conduct a prospective study for the evaluation of endocrine deficiency with aSAH. The investigators study patients 3, 6 and 12 month after aneurismal bleeding. Patients diagnosed with aSAH with a clinical grade of I-IV according to Hunt and Hess are included in the study. The investigators perform basal testing for the pituitary by measuring: TSH, LH, FSH, IGF-1, GH, prolactin and ACTH. For evaluation of the adrenal function the investigators perform an ACTH-stimulation test (Lindholm et al.). Subjects with evidence for adrenal or GH insufficiency are further analyzed by insulin-induced hypoglycemia testing (GH Research Society). In the neuropsychological examination, the investigators screen for verbal comprehension (Token Test, short form) and visual neglect (line bisection). Verbal and visual short term memory (digit and spatial span), visuospatial construction and figural memory (Rey Osterrieth Complex Figure Test), psychomotor speed, attention and concentration (Trail Making Test Part A and B, d2) as well as mental flexibility (word fluency) are assessed. Patients additionally fill out a questionnaire measuring actual depressive symptoms and anxiety (Hospital Anxiety and Depression Scale).

ELIGIBILITY:
Inclusion Criteria:

* aSAH grade I-IV Hunt und Hess
* bleeding CCT Fisher grade 3-4
* therapy within 48h after aSAH
* preoperative angiography as well as control angiography
* Glasgow Outcome Scale 4 to 5 after therapy

Exclusion Criteria:

* known intra-, peri- or suprasellar neoplasia
* preexisting hypopituitarism of any degree
* previous hormonal substitution
* previous radiation
* for the neuropsychological examination: difficulties with German language

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with aSAH with a clinical grade of I-IV according to Hunt and Hess are included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Estimated)
Dates: Start 2008-02; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
hypopituitarism of any degree | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsmedizin Mannheim, Mannheim, Baden-Wurttemberg, Germany

REFERENCES:
- [Background] Suarez JI, Tarr RW, Selman WR. Aneurysmal subarachnoid hemorrhage. N Engl J Med. 2006 Jan 26;354(4):387-96. doi: 10.1056/NEJMra052732. No abstract available. PMID 16436770
- [Background] Ogden JA, Mee EW, Henning M. A prospective study of impairment of cognition and memory and recovery after subarachnoid hemorrhage. Neurosurgery. 1993 Oct;33(4):572-86; discussion 586-7. doi: 10.1227/00006123-199310000-00004. PMID 8232796
- [Background] Anderson SW, Todd MM, Hindman BJ, Clarke WR, Torner JC, Tranel D, Yoo B, Weeks J, Manzel KW, Samra S. Effects of intraoperative hypothermia on neuropsychological outcomes after intracranial aneurysm surgery. Ann Neurol. 2006 Nov;60(5):518-527. doi: 10.1002/ana.21018. PMID 17120252
- [Background] Schneider HJ, Kreitschmann-Andermahr I, Ghigo E, Stalla GK, Agha A. Hypothalamopituitary dysfunction following traumatic brain injury and aneurysmal subarachnoid hemorrhage: a systematic review. JAMA. 2007 Sep 26;298(12):1429-38. doi: 10.1001/jama.298.12.1429. PMID 17895459
- [Background] Brabant G, Krogh Rasmussen A, Biller BM, Buchfelder M, Feldt-Rasmussen U, Forssmann K, Jonsson B, Koltowska-Haggstrom M, Maiter D, Saller B, Toogood A. Clinical implications of residual growth hormone (GH) response to provocative testing in adults with severe GH deficiency. J Clin Endocrinol Metab. 2007 Jul;92(7):2604-9. doi: 10.1210/jc.2007-0153. Epub 2007 May 8. PMID 17488801
- [Background] Lindholm J, Kehlet H. Re-evaluation of the clinical value of the 30 min ACTH test in assessing the hypothalamic-pituitary-adrenocortical function. Clin Endocrinol (Oxf). 1987 Jan;26(1):53-9. doi: 10.1111/j.1365-2265.1987.tb03638.x. PMID 3026692
- [Background] Growth Hormone Research Society. Consensus guidelines for the diagnosis and treatment of growth hormone (GH) deficiency in childhood and adolescence: summary statement of the GH Research Society. GH Research Society. J Clin Endocrinol Metab. 2000 Nov;85(11):3990-3. doi: 10.1210/jcem.85.11.6984. No abstract available. PMID 11095419